CLINICAL TRIAL: NCT04555369
Title: Study on the Efficacy of Chemotherapy for Metastatic Colorectal Cancer Evaluated by Circulating Tumor DNA
Brief Title: The Value of ctDNA on Chemotherapy Efficacy for mCRC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, MD,PhD, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: mCRC-ctDNA FUSCC
Record Dates: First submitted 2020-09-15; First posted 2020-09-18 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2020-09

CONDITIONS: Circulating Tumor DNA
MeSH Terms: interventions — Circulating Tumor DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ct-DNA (Experimental): The enrolled mCRC patients will perform ct-DNA testing to evaluate drug efficacy of chemotherapy, at the time of baseline and after the first cycle of chemotherapy.
  Interventions: Genetic: ct-DNA

INTERVENTIONS:
Genetic: ct-DNA — The enrolled mCRC patients will perform ct-DNA testing to evaluate drug efficacy of chemotherapy, at the time of baseline and after the first cycle of chemotherapy.
  Other Names: circulating tumor DNA

SUMMARY:
The study is designed to evaluate the value of ctDNA in predicting the drug efficacy of chemotherapy for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

aged ≥18 years with histologically or cytologically confirmed advanced colorectal adenocarcinoma Eastern Cooperative Oncology Group performance status of 0 to 2 life expectancy of ≥ 3 months at least one measurable metastatic lesion have adequate bone marrow, hepatic, and renal function

Exclusion Criteria:

patients with previous chronic inflammatory bowel disease, chronic diarrhea or recurrent bowel obstruction patients with symptomatic brain metastases active clinical severe infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 months
  the response rate predicted by ct-DNA

SECONDARY OUTCOMES:
Progression free survival | 2 months
Overall survival | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No